CLINICAL TRIAL: NCT01070108
Title: EARLY PREOPERATIVE ESCALATING DOSES OF KETAMINE ATTENUATE POSTOPERATIVE PAIN AND REDUCE MORPHINE CONSUMPTION IN HUMANS
Brief Title: Escalating Ketamine Doses and Pre-emption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Weinbroum Avraham, Tel Aviv Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ketamine
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2010-02

CONDITIONS: Postoperative Pain Management
Keywords: Preemption, ketamine, escalating, dose, pain, analgesia
MeSH Terms: conditions — Pain; Agnosia | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Set 1 (Active Comparator): group receiving one injection (25 mg) of ketamine (K1) intramuscularly (IM) at 3-4 hours before surgery or placebo (saline 0.9%, NS)
  Interventions: Drug: Ketamine
- set 2 (Active Comparator): 2nd set received ketamine at 11-12 hours (10 mg) and 3-4 hours (25 mg) before surgery (K2), with a corresponding NS group
  Interventions: Drug: ketamine
- set 3 (Active Comparator): 3rd set one group had ketamine injected IM 17-18, 11-12, and 3-4 hours before surgery (5, 10 and 25 mg, respectively) (K3), and the second group received NS
  Interventions: Drug: ketamine

INTERVENTIONS:
Drug: Ketamine — group receiving one injection (25 mg) of ketamine (K1) intramuscularly (IM) at 3-4 hours before surgery or placebo (saline 0.9%, NS)
  Arms: Set 1
Drug: ketamine — ketamine at 11-12 hours (10 mg) and 3-4 hours (25 mg) before surgery (K2), with a corresponding NS group
  Arms: Set 1; set 2
Drug: ketamine — ketamine injected IM 17-18, 11-12, and 3-4 hours before surgery (5, 10 and 25 mg, respectively) (K3), and the second group received NS

SUMMARY:
Ketamine affects postoperative pain when administered intravenously immediately before, during or at the end of surgical procedures. We assessed the effects of multiple and escalating doses of ketamine administered many hours before surgery on postoperative pain and analgesia consumption.

ELIGIBILITY:
Inclusion Criteria:

Consecutive patients, who were scheduled to undergo general or orthopedic oncologic surgery under general anesthesia

Exclusion Criteria:

1. allergy to opioids, ketamine or non-steroidal anti-inflammatory drugs (NSAIDs)
2. history of lasting chronic pain or psychiatric disorders or had used opioids or psychotropic drugs of any sort during the past two weeks
3. soldiers and pregnant women

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
postoperative pain | 48 hours

SECONDARY OUTCOMES:
opioid drug consumption | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel

REFERENCES:
- [Derived] Rakhman E, Shmain D, White I, Ekstein MP, Kollender Y, Chazan S, Dadia S, Bickels J, Amar E, Weinbroum AA. Repeated and escalating preoperative subanesthetic doses of ketamine for postoperative pain control in patients undergoing tumor resection: a randomized, placebo-controlled, double-blind trial. Clin Ther. 2011 Jul;33(7):863-73. doi: 10.1016/j.clinthera.2011.05.094. Epub 2011 Jul 1. PMID 21722959